CLINICAL TRIAL: NCT00005872
Title: Phase II Study of RFS 2000 in Relapsed NSCLC
Brief Title: Nitrocamptothecin in Treating Patients With Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067908; SUPERGEN-RFS2000-16; DFCI-99184
Record Dates: First submitted 2000-06-02; First posted 2004-04-12 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-09

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, time to progression and overall survival of patients with recurrent non-small cell lung cancer when treated with nitrocamptothecin. II. Assess the toxicities and pharmacokinetics of this regimen in these patients.

OUTLINE: Patients receive oral nitrocamptothecin daily on days 1-5. Treatment continues weekly in the absence of disease progression or unacceptable toxicity. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 20-55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent non-small cell lung cancer No more than one prior chemotherapy treatment Bidimensionally measurable disease No prior radiotherapy to target lesion OR Progression since prior radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL ALT/AST no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN in case of liver metastases) Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 50 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No uncontrolled serious medical or psychiatric illness

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy and recovered No prior camptothecin Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy and recovered Surgery: At least 2 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-05; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Show-Li Sun, MD, Study Chair — Astex Pharmaceuticals, Inc.
Locations (1):
- SuperGen, Incorporated, Dublin, California, United States